CLINICAL TRIAL: NCT05338684
Title: Role of the Radiologist in Management of Pulsatile Tinnitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mohab Mohammed (Other)
Responsible Party: Sponsor-Investigator, Mohab Mohammed, Role of the Radiologist in Management of Pulsatile tinnitus, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Radiology role in tinnitus
Record Dates: First submitted 2022-04-02; First posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Pulsatile Tinnitus (Diagnosis)
MeSH Terms: conditions — Tinnitus; Disease

STUDY DESIGN:
Intervention Model Description: patients diagnosed with pulsatile tinnitus clinically
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- diagnostic catheter intervention then therapeutic if indicated (Experimental)
  Interventions: Device: Colour doppler,MSCT,MRI

INTERVENTIONS:
Device: Colour doppler,MSCT,MRI — ultrasound/color duplex at Jugular veins & carotid and vertebral arteries first ,then MSCT/CTA mainly with relation of neck & Bain arteries to the bone of the skull in 6 mm cuts and/or MRI/MRA/MRV by standardized multi-parametric MR protocol will be implemented for all patients. All sequences will be acquired on a 1.5T MR scanner.

SUMMARY:
The aim of this study is to detect the role of interventional radiology in management of Pulsatile tinnitus and to detect the best imaging modality for Diagnosis.

DETAILED DESCRIPTION:
Tinnitus is a broad and complex subject concerning a symptom rather than a syndrome or a disease (1 ),New studies indicate that prevalence of tinnitus is 14.5% among those less than 40 years old and 17.5 - 35% among age over 40 years Old( 2-3 ). Vascular tinnitus causes are multiple , Arterial causes like Atherosclerosis , Fibromuscular dysplasia or Dissection of the carotid or vertebral artery , Arteriovenous causes like Cerebral head and neck arteriovenous malformation , Dural arteriovenous fistula and Carotid cavernous fistula Venous like Systemic diseases with hyperdynamic circulation . Chronic anemia, pregnancy, thyrotoxicosis , Idiopathic intracranial hypertension and Dural venous sinus stenosis , Tumors also like Paraganglioma which Some authors believe that para-gangliomas are the most common cause of vascular tinnitus and Vascular metastasis And other Miscellaneous Causes like Paget's disease m Otosclerosis or Otomastoiditis , but others see dural arteriovenous fistula (AVF) ,idiopathicvenous tinnitus, or idiopathic intracranial hypertension the most common causes. (4 - 9) , Also One of the Most important Arterial causes is Atherosclerosis , Atherosclerotic plaques ma produce turbulence of carotid flow and occasionally cause pulsatile tinnitus (10 ) , FMD ( Fibromuscular Dysplasia ) seen in 0.5% to0.6% of carotid angiograms and autopsies, is the second most common cause of extracranial carotid narrowing (11) information obtained from both CT and MRI is complementary In some casesThe angiographic findings may include luminal stenosis, abrupt reconstitution of the lumen, dissecting aneurysm, intimal flap, slow flow, occlusion, and distal emboli (12-15)

ELIGIBILITY:
Inclusion Criteria:

* Patients with pulsatile tinnitus of unknown origin referred by a physician to diagnostic radiology to be assessed by imaging will be included in the study.
* Patient's with clinical diagnosed pulsatile tinnitus.
* patient refused surgical intervention.

Exclusion Criteria:

* History of allergy to the contrast media , Contraindication to MRI and Refusal to sign a consent
* Pregnant women
* patients with atherosclerosis cause only or vascular loop more than 50% in internal auditory canal

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-17 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Manage pulsatile tinnitus with catheter angiography to all vascular lesion | Baseline
  Manage pulsatile tinnitus causes with no indication for surgical intervention or prolonged and follow up and detect reported cases with pulsatile tinnitus could be managed by therapeutic angiography rather than other invasive surgical maneuver or Medical treatment

SECONDARY OUTCOMES:
To assess the accuracy of best imaging modality to diagnose pulsatile tinnitus . | Baseline
  Detect accurate cause of pulsatile tinnitus and the best imaging for diagnosis with measurement of the percentage of indicated patient for therapeutic angiography rather than surgical intervention or follow up with medical treatment .

REFERENCES:
- [Background] Noell CA, Meyerhoff WL. Tinnitus. Diagnosis and treatment of this elusive symptom. Geriatrics. 2003 Feb;58(2):28-34. PMID 12596495
- [Background] Heller AJ. Classification and epidemiology of tinnitus. Otolaryngol Clin North Am. 2003 Apr;36(2):239-48. doi: 10.1016/s0030-6665(02)00160-3. PMID 12856294
- [Background] Mehanna R, Shaltoni H, Morsi H, Mawad M. Endovascular treatment of sigmoid sinus aneurysm presenting as devastating pulsatile tinnitus. A case report and review of literature. Interv Neuroradiol. 2010 Dec;16(4):451-4. doi: 10.1177/159101991001600413. Epub 2010 Dec 17. PMID 21162777
- [Background] Schleuning A. Neurotologic evaluation of subjective idiopathic tinnitus. J Laryngol Otol Suppl. 1981;(4):99-101. No abstract available. PMID 6946175
- [Background] Dietz RR, Davis WL, Harnsberger HR, Jacobs JM, Blatter DD. MR imaging and MR angiography in the evaluation of pulsatile tinnitus. AJNR Am J Neuroradiol. 1994 May;15(5):879-89. PMID 8059655
- [Background] George B, Reizine D, Laurian C, Riche MC, Merland JJ. Tinnitus of venous origin. Surgical treatment by the ligation of the jugular vein and lateral sinus jugular vein anastomosis. J Neuroradiol. 1983;10(1):23-30. No abstract available. English, French. PMID 6864262
- [Background] Sismanis A. Pulsatile tinnitus. A 15-year experience. Am J Otol. 1998 Jul;19(4):472-7. PMID 9661757
- [Background] Sismanis A. Pulsatile tinnitus. Otolaryngol Clin North Am. 2003 Apr;36(2):389-402, viii. doi: 10.1016/s0030-6665(02)00169-x. PMID 12856306
- [Background] Waldvogel D, Mattle HP, Sturzenegger M, Schroth G. Pulsatile tinnitus--a review of 84 patients. J Neurol. 1998 Mar;245(3):137-42. doi: 10.1007/s004150050193. PMID 9553842
- [Background] Sandok BA, Whisnant JP, Furlan AJ, Mickell JL. Carotid artery bruits: prevalence survey and differential diagnosis. Mayo Clin Proc. 1982 Apr;57(4):227-30. PMID 7070118
- [Background] Corrin LS, Sandok BA, Houser OW. Cerebral ischemic events in patients with carotid artery fibromuscular dysplasia. Arch Neurol. 1981 Oct;38(10):616-8. doi: 10.1001/archneur.1981.00510100044005. PMID 7295104
- [Background] Gelbert F, Assouline E, Hodes JE, Reizine D, Woimant F, George B, Hagueneau M, Merland JJ. MRI in spontaneous dissection of vertebral and carotid arteries. 15 cases studied at 0.5 tesla. Neuroradiology. 1991;33(2):111-3. doi: 10.1007/BF00588245. PMID 2046892